CLINICAL TRIAL: NCT01961635
Title: Healing Response if Peri-implant Tissues to Different Abutment Materials - Double-blinded Randomized Clinical Trial
Brief Title: Healing of Bone/Soft Tissue to Different Abutment Biomaterials and the Impact on Marginal Bone Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Implantology Institute (Other)
Responsible Party: Principal Investigator, Andre Chen, Msc, Implantology Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: II-01
Record Dates: First submitted 2013-10-06; First posted 2013-10-11 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Bone Loss; Inflammation
Keywords: Dental Implants; Zirconia Abutments; Titanium abutments; Acrylic abutments; Gingival Healing; Inflammation; Bone loss
MeSH Terms: conditions — Bone Diseases, Metabolic; Inflammation | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zirconia Abutments (Experimental): Place zirconia one-time one-abutment in subcrestal platform-switch dental implants on the day of implant installation, torque 20 n/cm2
  Interventions: Device: dental implants; Device: Zirconia abutments; Procedure: Subcrestal; Device: platform-switch; Procedure: one-time one-abutment; Procedure: Torque 20 n/cm2
- Titanium Abutments (Experimental): Place titanium one-time one-abutment in subcrestal platform-switch dental implants on the day of implant installation, torque 20 n/cm2
  Interventions: Device: dental implants; Device: Titanium Abutments; Procedure: Subcrestal; Device: platform-switch; Procedure: one-time one-abutment; Procedure: Torque 20 n/cm2
- Cad-Cam Acrylic abutments (Experimental): Place cad-cam acrylic one-time one-abutment in subcrestal platform-switch dental implants on the day of implant installation, torque 20 n/cm2
  Interventions: Device: dental implants; Device: cad-cam acrylic abutments; Procedure: Subcrestal; Device: platform-switch; Procedure: one-time one-abutment; Procedure: Torque 20 n/cm2

INTERVENTIONS:
Device: dental implants — place implant according fabricant guidelines, 2mm sub-crestally
  Other Names: T3 - Biomet 3I Implants; Platform-Switch 4.1; Abutment Diameter 3.25
Device: Zirconia abutments — place zirconia abutment on the day of implant placement
  Other Names: Zirconia cad-cam abutment; 3.25 Abutment connection
  Arms: Zirconia Abutments
Device: Titanium Abutments — place titanium abutment on the day of implant placement
  Other Names: Titanium Encode - biomet 3I Implants; 3,25 abutment connection
  Arms: Titanium Abutments
Device: cad-cam acrylic abutments — place cad-cam acrylic abutment on the day of implant placement
  Other Names: Cad-cam acrylic abutment; 3.25 platform
  Arms: Cad-Cam Acrylic abutments
Procedure: Subcrestal — place implant 2mm below crestal bone
Device: platform-switch — abutment platform is narrow than implant diameter
Procedure: one-time one-abutment — place the final abutment on the day of surgery and not remove it
  Other Names: one time abutment; final abutment on the day of surgery
Procedure: Torque 20 n/cm2 — the amount of torque applied to the abutment
  Other Names: manual torque

SUMMARY:
In patients that require a dental implant, does zirconia compared to titanium, or cad-cam acrylic abutments, provide less inflammation, marginal bone loss or infection during the osseointegration period ?

DETAILED DESCRIPTION:
Place dental Implants and zirconia, titanium, acrylic or cad-cam acrylic abutments, torque to 20 n/cm2 Evaluate Changes in inflammatory levels from T0 (baseline) to T7-12 weeks (measure intermediate points at T0 (baseline),,T1-8 Weeks and T2-12 weeks) Also evaluate outcomes marginal bone loss, gingival height levels and osseointegration

ELIGIBILITY:
Inclusion Criteria:

* Single unit implant rehabilitation
* Maxilla and mandible
* Must accept treatment plan
* Must sign informed consent
* dental extraction performed at least 3 month prior
* Must have at least 6 mm of residual bone
* Absence of oral lesions
* keratinized tissue must be present

Exclusion Criteria:

* If smoking and/or other drug addiction is present
* If local anesthetic allergy is present
* Patient subjected to chemical or radiotherapy
* if Hepatic disease is present
* If immunodepression is present
* If Pregnancy is present
* If Diabetes is present
* If Heart disease is present

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Gingival Inflammatory Changes from baseline to 12 weeks | Measure - T0 Implant installation T1- 1week post-surgery T2-two weeks T3-3weeks T4-4weeks T5-6weeks T6-8weeks T7-12 weeks
  measure the amount of cytokines and interleukines (interleukin-8 (IL-8), macrophage inflammatory protein-1 (MIP-1 beta), interleukin-1 (IL-1 beta), interleukin-6 (IL-6), matrix metalloproteinase-8 (MMP-8) and matrix metalloproteinase-9 (MMP-9), metallopeptidase inhibitor 1 (TIMP-1), vascular endothelial growth factor (VEGF)), around different implant abutment materials, zirconia,titanium, acrylic, and cad-cam acrylic

SECONDARY OUTCOMES:
Marginal Bone Loss | measured at 12 weeks post-implant installation
  Parallel periapical standardized radiographs to measure bone position in relation to implant platform, in zirconia,titanium, acrylic, and cad-cam acrylic
Gingival height | 12 weeks post-implant installation
  measure with periodontal probe distance from implant platform to the most coronal point of gingival margin mesial, distal, buccal and lingual,in zirconia,titanium, acrylic, and cad-cam acrylic
Osseointegration | 12 weeks post-implant installation
  compare survival rate of dental implants rehabilitated with zirconia,titanium, acrylic, and cad-cam acrylic abutments
Height from gingiva to abutment | 12 weeks post implant installation
  height from gingival margin to most coronal point of the abutment in zirconia, titanium, acrylic and acrylic cad-cam abutments

CONTACTS AND LOCATIONS:
Overall Officials: João Caramês, Phd, Principal Investigator — Faculdade de Medicina Dentária de Lisboa; André Chen Chen, Msc, Study Director — Faculdade de Medicina Dentária de Lisboa; Elena Cervino, Msc, Study Chair — Implantology Institute; Helena Francisco, Phd, Study Chair — Faculdade de Medicina Dentária de Lisboa
Locations (1):
- Faculdade de Medicina Dentária de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided